CLINICAL TRIAL: NCT02667158
Title: A Survey Study to Evaluate the Relation Between Doctor/Pharmacy Shopping and Outcomes Suggestive of Misuse, Abuse and/or Diversion
Brief Title: A Survey to Eval the Relation Between Doctor/Pharmacy Shopping and Outcomes Suggestive of Misuse, Abuse and/or Diversion
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-9; 3033-9 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- No shopping behavior: Patients will be grouped into one of the categories based on the most recent 18 months of data available at the time the patient sample is identified
  Interventions: Other: Survey to Eval Relation between Shopping and Misuse, Abuse
- Minimal shopping behavior: Patients will be grouped into one of the categories based on the most recent 18 months of data available at the time the patient sample is identified
  Interventions: Other: Survey to Eval Relation between Shopping and Misuse, Abuse
- Marked shopping behavior: Patients will be grouped into one of the categories based on the most recent 18 months of data available at the time the patient sample is identified
  Interventions: Other: Survey to Eval Relation between Shopping and Misuse, Abuse
- Extensive shopping behavior: Patients will be grouped into one of the categories based on the most recent 18 months of data available at the time the patient sample is identified
  Interventions: Other: Survey to Eval Relation between Shopping and Misuse, Abuse

INTERVENTIONS:
Other: Survey to Eval Relation between Shopping and Misuse, Abuse — A Survey Study to Evaluate the Relation Between Doctor/Pharmacy Shopping and Outcomes Suggestive of Misuse, Abuse and/or Diversion

SUMMARY:
To evaluate the reasons patients go to more than one prescriber or more than one pharmacy to obtain prescriptions opioids and assess whether the percentage of patients reporting misuse, abuse and/or diversion increases across defined categories of doctor/pharmacy shopping as defined in Study 4A.

DETAILED DESCRIPTION:
Based on a review of the literature, the Food and Drug Administration (FDA) concluded that more data are needed regarding the serious risks of misuse, abuse, addiction, overdose, and death associated with the long-term use of extended release/long acting (ER/LA) opioid analgesics. Thus, the FDA is requiring that ER/LA opioid analgesic drug sponsors conduct post-marketing studies to assess these risks. The four observational post-marketing requirement (PMR) studies are labeled Study #2065-1, Study #2065-2, Study #2065-3, and Study #2065-4.

The objective of PMR Study #2065-4 is to define and validate doctor/pharmacy shopping as outcomes suggestive of misuse, diversion, abuse and/or addiction.

Study #2065-4 consists of three sub-studies, Study 4A, Study 4B, and Study 4C. In the current study (#2065-4 sub-study, Study 4B), the association between doctor/pharmacy shopping behavior and misuse, diversion and abuse will be assessed by surveying patients within the a priori defined four categories of shopping behaviors. The four categories of shopping behaviors identified and defined in Study 4A will be applied to Study 4B. Asking patients directly about their behaviors related to misuse and abuse will provide us with the patient's perspective that is unavailable in Study 4A. Surveying patients regarding misuse and abuse requires the use of an instrument that has undergone a validation process to ensure that misuse and abuse are being measured. Study 4B will utilize the Prescription Opioid Misuse and Abuse Questionnaire (POMAQ) that will be validated in PMR Study #2065-2A. An administrative claims database will be used to identify the eligible patient population using their pharmacy claims for immediate release (IR) or ER/LA opioid analgesics to determine the number of prescribers and number of pharmacies they visit. Consenting patients will be asked to complete an online survey that includes the POMAQ to self-report their behaviors of misuse, abuse and/or diversion. It is hypothesized that as the likelihood of doctor/pharmacy shopping behavior increases the risk of misuse, abuse and/or diversion.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria:

1. At least two pharmacy claims for any IR or ER/LA opioid analgesic in the most recent 18 months of claims data.
2. Based on claims for the most recent 18 months of data, meet classification criteria for one of the four a priori defined doctor/pharmacy shopping categories.
3. Currently active, commercially-insured, survey eligible with medical and pharmacy benefits with a health plan included in the HealthCore Integrated Research Database (HIRD) at the time the sample list is extracted.
4. At least 18 years of age as of the date of the first IR or ER/LA opioid dispensing in the most recent 18 months of claims data.
5. A telephone number or address known to HealthCore.

Exclusion Criteria:

1. Patients who appear on the HealthCore "Do-not-call" list.
2. Patients with a known history of abuse
3. Patients who do not indicate that they have read about all pertinent aspects of the study and agree to participate.
4. Patients who fail to validate their name and/or date of birth
5. Patients who are unable to understand the survey questions as designed (e.g., non-English speaking, etc.).
6. Patients who fail other study-specific screening questions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (18 years of age or older) identified from the HealthCore Integrated Research Database (HIRD) with at least two pharmacy claims for any IR or ER/LA opioid analgesic in the most recent 18 months of claims data
Sampling Method: Probability Sample
Enrollment: 1085 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Self-reported reasons that patients go to more than one prescriber or more than one pharmacy, stratified by doctor/pharmacy shopping categories | Day 1, based upon single patient survey completed online or via telephone
Responses suggestive of misuse and/or abuse on the POMAQ. | Day 1, based upon single patient survey completed online or via telephone

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Cepeda, MD, PhD, Study Chair — Janssen Research & Development, LLC